CLINICAL TRIAL: NCT00498914
Title: A Phase II Multicenter, Open-Label Study of YM155 in Refractory Diffuse Large B-Cell Lymphoma (DLBCL) Subjects
Brief Title: Study of YM155 in Refractory Diffuse Large B-cell Lymphoma (DLBCL) Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility boundary at interim analysis not met
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 155-CL-009; Eudra CT 2006-002584-70
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-08

CONDITIONS: Lymphoma, Large-Cell, Diffuse; Lymphoma, B-Cell Refractory
Keywords: Lymphoma, Large-Cell, Diffuse; Lymphoma, B-Cell; YM155; Treatment outcomes; Refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Lymphoma, B-Cell | interventions — sepantronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: YM155

INTERVENTIONS:
Drug: YM155 — Continuous IV infusion

SUMMARY:
A study in subjects with a type of B cell lymphoma (DLBCL)to evaluate the response rate, efficacy, safety and tolerability of YM155

DETAILED DESCRIPTION:
1 arm (Active), Phase 2 Study to evaluate response rate, efficacy, safety and tolerability of YM155

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older
* Histologically confirmed primary DLBCL of any stage
* Refractory to the last treatment regimen
* Previously treated with the following treatment regimens:
* Anthracycline-based combination chemotherapy with rituximab
* Second-line combination chemotherapy
* Autologous BMT if the subject was eligible and did not refuse the procedure
* At least one measurable lesion defined as > 1.5 cm in the longest diameter
* No known central nervous system involvement
* ECOG performance status < 2
* Life expectancy > 12 weeks
* If female, non-pregnant and non-lactating
* IRB-approved consent and HIPAA Authorization

Exclusion Criteria:

* Transformed, composite or discordant lymphoma
* Therapy for lymphoma within 21 days prior to the first dose of YM155
* Within 4 weeks of the screening FDG-PET scan, receipt of the following:
* Radiation therapy
* Surgical procedures (except biopsies and central catheter / port placement)
* Active infection (bloodstream or deep tissue)
* Inadequate marrow, hepatic and/or renal function
* Serum creatinine > 1.5 x ULN or calculated serum creatinine clearance < 60 mL/min
* Absolute Neutrophil Count (ANC) < 750/mm3
* Platelet < 50,000/mm3
* Alanine Transaminase (ALT) and Aspartate Transaminase (AST) > 2.5 x ULN; > 5 x ULN if secondary to liver metastases
* Treated with > 3 prior treatment regimens. The following should be considered:
* Planned maintenance therapy should be considered as part of the previous treatment regimen
* Any preparative treatment (salvage chemotherapy, high-dose chemotherapy, radiation therapy, etc.) should be included with the autologous BMT or PBSCT as one treatment
* Prior allogeneic BMT or PBSCT
* Previously treated with YM155
* Other investigational therapy or procedures within 28 days
* Known HIV, hepatitis B surface antigen, or hepatitis C antibody
* Other malignancy requiring treatment within 2 years
* Significant and/or uncontrolled cardiac, renal, hepatic, or other systemic disorders or significant psychological conditions that in the Investigator's judgment would jeopardize subject enrollment or compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 15 treatment cycles

SECONDARY OUTCOMES:
Safety, efficacy, pharmacokinetics, and tolerability | 15 treatment cycles

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (22):
- United States (12):
  - Beverly Hills, California
  - Palo Alto, California
  - Aurora, Colorado
  - Miami, Florida
  - Atlanta, Georgia
  - Shreveport, Louisiana
  - St Louis, Missouri
  - Winston-Salem, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - San Antonio, Texas
- Ottawa, Ontario, Canada
- France (7):
  - Bordeaux
  - Montpellier
  - Nantes
  - Nice
  - Poitiers
  - Rouen
  - Tours
- Spain (2):
  - Barcelona
  - Madrid